CLINICAL TRIAL: NCT03332901
Title: To Monitor the Effect on the Laparoscopic Pneumoperitoneum of Gastroesophageal Function During Anesthesia
Brief Title: Gastroesophageal Function During Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201708035RINA
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Gastroesophageal Function During General Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: this is an observational study, no intervention required — this is an observational study, no intervention required

SUMMARY:
General anesthesia may predispose patients to aspiration of gastroesophageal contents because of depression of protective reflexes during loss of consciousness. The laparoscopy would increase the intra-abdominal pressure, which is regarded as a predisposing factor of gastroesophageal reflux during the anesthesia. The lower esophageal sphincter is the important physiological mechanisms that prevent regurgitation and aspiration. However, the change of LES pressure and gastroesophageal reflux before and after laparoscopic physiological condition is still unknown because the prospective evaluation of gastroesophageal function in human is limited. In addition, the relationship between the change of intra-abdominal pressure and the LES pressure were still unknown, too. In this study, we aimed to observe the changes of gastroesophgeal function parameters by esophageal manometry, pH impedance, and intra-abdominal pressure measured by AbViser ®AutoValve®IAP Monitoring Device before and after laparoscopic condition.

DETAILED DESCRIPTION:
Background: General anesthesia may predispose patients to aspiration of gastroesophageal contents because of depression of protective reflexes during loss of consciousness. The laparoscopy would increase the intra-abdominal pressure, which is regarded as a predisposing factor of gastroesophageal reflux during the anesthesia. The lower esophageal sphincter is the important physiological mechanisms that prevent regurgitation and aspiration. However, the change of LES pressure and gastroesophageal reflux before and after laparoscopic physiological condition is still unknown because the prospective evaluation of gastroesophageal function in human is limited. In addition, the relationship between the change of intra-abdominal pressure and the LES pressure were still unknown, too.

The esophageal manometry has pressure sensor to measure the LES pressure. The AbViser ®AutoValve®IAP Monitoring Device is a sterile non-invasive disposable monitoring device, that is routinely used to measure intra-abdominal pressure (IAP) in the intensive care unit. Therefore, application of esophageal manometry and pH impedance via second-generation SADs may help to detect gastroesophageal functional change and ongoing gastroesophageal regurgitation during perioperative period. We also used the AbViser ®AutoValve®IAP Monitoring Device to monitor the change of IAP before and after laparoscopic condition. In this study, we aimed to observe the changes of gastroesophgeal function parameters by esophageal manometry and intra-abdominal pressure measured by AbViser ®AutoValve®IAP Monitoring Device before and after laparoscopic condition.

Objectives: we aimed to observe the changes of gastroesophgeal function parameters by esophageal manometry, pH impedance, and intra-abdominal pressure measured by AbViser ®AutoValve®IAP Monitoring Device before and after laparoscopic condition.

Patients and methods: Consecutive patients who will receive scheduled laparoscopic surgery under general anesthesia and aged >= 20 will be enrolled. All subjects provide basic demographic data and fill in standard symptom questionnaire for evaluation of baseline upper gastrointestinal symptoms. After induction, the endotracheal tube (ETT) will be inserted to establish airway. Then, the esophageal manometry would be inserted to monitor the LES, and the AbViser ®AutoValve®IAP Monitoring Device will be inserted to monitor the IAP before and after the laparoscopic condition. After the surgery and removal of ETT, the patients will be followed for the oxygen saturation, sore throat or hoarseness in the postoperative care unit, as well as the possible complications.

Expected result: We will observe the changes of LES function, gastroesophageal reflux and the relationship between the IAP and the LES function before and after the laparoscopic condition.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who will receive scheduled laparoscopic surgery under general anesthesia 2. Aged from 20-80 years old

Exclusion Criteria:

- 1. Major systemic disease, such as congestive heart failure, liver cirrhosis, end stage renal disease and malignancy.

2. Patients who have the risk of difficult ventilation or intubation. 3. pregnant women 4. coagulopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will receive scheduled laparoscopic surgery under general anesthesia; Aged from 20-80 years old
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-03-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
lower esophaegal sphincter pressure | during the anesthesia

SECONDARY OUTCOMES:
episodes of reflux | duirng the anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Jung Cheng, MD,PhD, Principal Investigator — anesthesiology of department, National Taiwan university hospital
Locations (1):
- Ya-Jung, Cheng, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Lai CJ, Chang WC, Huang CH, Liu CM, Lo YC, Cheng YJ. Detecting intraoperative gastric regurgitation by using preattached esophageal multichannel intraluminal impedance and pH monitoring on a solid-state manometry: a case series study. J Clin Monit Comput. 2020 Aug;34(4):853-859. doi: 10.1007/s10877-019-00380-2. Epub 2019 Aug 29. PMID 31468255